CLINICAL TRIAL: NCT02541981
Title: Natural Course for Renal Function After Heart Transplantation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201507087RIND
Record Dates: First submitted 2015-08-31; First posted 2015-09-04 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Creatinine Clearance Quantitative Trait Locus
Keywords: Heart transplant; renal insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The outcome of heart transplantation has improved by years. The renal dysfunction is a major complication after heart transplantation.The natural course of renal function following orthotopic heart transplant is not clear in Taiwan. A retrospective study was conducted on patients who received a heart transplant at National Taiwan University Hospital between 1987 and 2015.

DETAILED DESCRIPTION:
The investigators conducted a retrospective cohort study of patients who received a first heart transplant at the NTUH(Taiwan) between 1987 and 2015 . Clinical data were obtained and a retrospective chart review, and were collected up to 10 years .

Data was collected from medical records and the heart transplant electronic database including: demographic parameters such as age and gender; etiology of heart failure; the presence of any of the following comorbidities: history of smoking, diabetes, hypertension, peripheral vascular disease and previous sternotomy; pre-transplant cholesterol levels; the use of any of the following pretransplant hemodynamic support measures:intravenous inotropes, intra-aortic balloon pump and ventricular assist device;creatinine levels; listing status according to the UNOS classification; waiting time; heart ischemic time;immunosuppression drug levels(cyclosporine,prograft or certican) and development of end stage renal disease requiring onset of dialysis therapy.

Creatinine levels and GFRwere collected before transplantation and then the closest level to every month after heart transplant.

The clinical outcomes of interest analyzed in this study included the development of post-transplant end stage renal disease and death.

ELIGIBILITY:
This study included patients with a first HTx performed at NTUH between1987 and 2015.

Patients were excluded if their first HTx was a combined transplant involving a KTx, they had renal replacement therapy prior to their HTx.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: heart transplantation
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Natural course for renal function (ex blood creatine leveal ,eGFR) after heart transplantation | patients who received a first heart transplant at the NTUH(Taiwan) between 1987 and 2015
  the outcome measure is assessed up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Chen Cheryl Chia-Hui, PHD, Principal Investigator — Professor , School of Nursing, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan